CLINICAL TRIAL: NCT06811324
Title: The Effects of Tirzepatide Use on Muscle and Vascular Function Among Obese Older Adults
Brief Title: Effects of Tirzepatide on Muscle and Vascular Health in Obese Older Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001208
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Obesity Prevention; Sarcopenia in Elderly; Cardiovascular Function; GLP - 1; Weight Loss
Keywords: Tirzepatide; GLP-1; Obesity; Sarcopenia; Cardiovascular Function
MeSH Terms: conditions — Weight Loss; Obesity; Sarcopenia | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirzepatide (Experimental): Tirzepatide self-administered once weekly by subcutaneous injection
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Once weekly tirzepatide starting at 2.5 mg/weekly, with dose escalation monthly by 2.5 mg to a target dose of 10 mg/weekly or maximum tolerated
  Other Names: Zepbound, LY3298176

SUMMARY:
Obesity and type 2 diabetes mellitus (T2DM) represent major public health concerns in the aging community. Tirzepatide, a novel dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 (GLP-1) receptor agonist recently approved for the treatment of T2DM and obesity has been shown to be effective at reducing weight, improving markers of T2DM control, and improving cardiovascular health. Utilization of tirzepatide among older adults has been on the rise since FDA approval was issued, however the effects of tirzepatide use on functional outcomes in older adults with obesity are not well established. Recent studies show that weight loss caused by tirzepatide may be driven by substantial loss of lean muscle mass, which may contribute to weakness and frailty, particularly among older adults. The proposed pilot study aims to evaluate how treatment with tirzepatide for 6 months affects muscle mass and function among older adults, and if changes in muscle mass are linked to changes in functional status over the same time period.

DETAILED DESCRIPTION:
This study is a pilot, single-arm, open-label clinical trial to evaluate the effects of Tirzepatide on muscle mass, strength, and vascular health among older adults with obesity. This study is set in South Texas, where rates of obesity and related health issues, including type 2 diabetes and cardiovascular conditions, exceed national averages and where aging-related diseases are on the rise. Tirzepatide is a new FDA approved medication that promotes weight loss and improves health by targeting specific pathways in the body. While it has been shown to be effective in managing weight and blood sugar levels, there is less information about the kind of weight loss it induces, and how weight loss impacts measures of muscle mass, strength and mobility. This is especially concerning for older adults, as losing muscle mass can lead to weakness, falls, and disability.

ELIGIBILITY:
Inclusion Criteria

* Men and postmenopausal women aged 50 years or older.
* Body Mass Index (BMI) ≥30 kg/m².
* Untreated HbA1c <6.5% at baseline.
* Willingness and ability to comply with all study procedures, including fasting requirements for certain visits.
* Able to provide informed consent and participate in all study assessments.

Exclusion Criteria

* Active diagnosis of type 2 diabetes mellitus (T2DM), defined by active use of glucose-lowering medications or hemoglobin A1c ≥ 6.5%.
* Body Mass Index (BMI) ≥ 40 kg/m².
* Moderate to severe gastroesophageal reflux disease based on patient history.
* Inability to comply with the treatment protocol or to understand the consent form.
* Chronic Kidney Disease (CKD) Stage 4.
* Aspartate aminotransferase (AST) > 33 U/L or alanine aminotransferase (ALT) > 36 U/L.
* Active pregnancy.
* Personal or family history of medullary thyroid carcinoma.
* Personal or family history of multiple endocrine neoplasia type 2 syndrome.
* Personal history of gastroparesis.
* Personal history of diabetic retinopathy.
* Known serious hypersensitivity, including anaphylaxis and angioedema, to Tirzepatide or any of its excipients.
* Known serious hypersensitivity, including anaphylaxis and angioedema, to any GLP-1 receptor agonist class of therapies.
* Concomitant treatment with GLP-1 receptor agonist therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Appendicular lean muscle mass | 6 months
  Appendicular lean muscle mass assessed at baseline and at 6-month follow-up by dual-energy X-ray absorptiometry (DEXA)
Muscle Strength | 6 months
  Muscle strength assessed by isokinetic and isometric testing using Biodex dynamometry at baseline and at 6-month follow-up.
Lower Extremity Functional Capacity | 6 months
  Functional capacity will be measured using the 6-minute walk test (6MWT) at baseline and 6-month follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Shreya Rao, MD, MPH, Principal Investigator — The University of Texas Health Science Center at San Antonio; Elena Volpi, MD, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Tiffany Cortes, MD, Study Director — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported will be available in accordance with ICMJE policy.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 1 year after the end of the trial and publication of the primary outcomes, and will be available for 24 months.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposals. Proposals should be directed to the principal investigators. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Marx N, Husain M, Lehrke M, Verma S, Sattar N. GLP-1 Receptor Agonists for the Reduction of Atherosclerotic Cardiovascular Risk in Patients With Type 2 Diabetes. Circulation. 2022 Dec 13;146(24):1882-1894. doi: 10.1161/CIRCULATIONAHA.122.059595. Epub 2022 Dec 12. PMID 36508493
- [Background] Clark RV, Walker AC, O'Connor-Semmes RL, Leonard MS, Miller RR, Stimpson SA, Turner SM, Ravussin E, Cefalu WT, Hellerstein MK, Evans WJ. Total body skeletal muscle mass: estimation by creatine (methyl-d3) dilution in humans. J Appl Physiol (1985). 2014 Jun 15;116(12):1605-13. doi: 10.1152/japplphysiol.00045.2014. Epub 2014 Apr 24. PMID 24764133
- [Background] Colleluori G, Villareal DT. Aging, obesity, sarcopenia and the effect of diet and exercise intervention. Exp Gerontol. 2021 Nov;155:111561. doi: 10.1016/j.exger.2021.111561. Epub 2021 Sep 23. PMID 34562568
- [Background] Wilkinson DJ, Piasecki M, Atherton PJ. The age-related loss of skeletal muscle mass and function: Measurement and physiology of muscle fibre atrophy and muscle fibre loss in humans. Ageing Res Rev. 2018 Nov;47:123-132. doi: 10.1016/j.arr.2018.07.005. Epub 2018 Jul 23. PMID 30048806
- [Background] Wadden TA, Chao AM, Machineni S, Kushner R, Ard J, Srivastava G, Halpern B, Zhang S, Chen J, Bunck MC, Ahmad NN, Forrester T. Tirzepatide after intensive lifestyle intervention in adults with overweight or obesity: the SURMOUNT-3 phase 3 trial. Nat Med. 2023 Nov;29(11):2909-2918. doi: 10.1038/s41591-023-02597-w. Epub 2023 Oct 15. PMID 37840095
- [Background] Conte C, Hall KD, Klein S. Is Weight Loss-Induced Muscle Mass Loss Clinically Relevant? JAMA. 2024 Jul 2;332(1):9-10. doi: 10.1001/jama.2024.6586. PMID 38829659
- [Background] Frias JP, Davies MJ, Rosenstock J, Perez Manghi FC, Fernandez Lando L, Bergman BK, Liu B, Cui X, Brown K; SURPASS-2 Investigators. Tirzepatide versus Semaglutide Once Weekly in Patients with Type 2 Diabetes. N Engl J Med. 2021 Aug 5;385(6):503-515. doi: 10.1056/NEJMoa2107519. Epub 2021 Jun 25. PMID 34170647
- [Background] Kaneko S. Tirzepatide: A Novel, Once-weekly Dual GIP and GLP-1 Receptor Agonist for the Treatment of Type 2 Diabetes. touchREV Endocrinol. 2022 Jun;18(1):10-19. doi: 10.17925/EE.2022.18.1.10. Epub 2022 Jun 16. PMID 35949358
- [Background] Koyama AK, McKeever Bullard K, Xu F, Onufrak S, Jackson SL, Saelee R, Miyamoto Y, Pavkov ME. Prevalence of Cardiometabolic Diseases Among Racial and Ethnic Subgroups in Adults - Behavioral Risk Factor Surveillance System, United States, 2013-2021. MMWR Morb Mortal Wkly Rep. 2024 Jan 25;73(3):51-56. doi: 10.15585/mmwr.mm7303a1. PMID 38271277
- [Background] Prado CM, Phillips SM, Gonzalez MC, Heymsfield SB. Muscle matters: the effects of medically induced weight loss on skeletal muscle. Lancet Diabetes Endocrinol. 2024 Nov;12(11):785-787. doi: 10.1016/S2213-8587(24)00272-9. Epub 2024 Sep 9. No abstract available. PMID 39265590
- [Background] Neeland IJ, Linge J, Birkenfeld AL. Changes in lean body mass with glucagon-like peptide-1-based therapies and mitigation strategies. Diabetes Obes Metab. 2024 Sep;26 Suppl 4:16-27. doi: 10.1111/dom.15728. Epub 2024 Jun 27. PMID 38937282
- [Background] Larsson L, Degens H, Li M, Salviati L, Lee YI, Thompson W, Kirkland JL, Sandri M. Sarcopenia: Aging-Related Loss of Muscle Mass and Function. Physiol Rev. 2019 Jan 1;99(1):427-511. doi: 10.1152/physrev.00061.2017. PMID 30427277
- [Background] Eberly LA, Yang L, Essien UR, Eneanya ND, Julien HM, Luo J, Nathan AS, Khatana SAM, Dayoub EJ, Fanaroff AC, Giri J, Groeneveld PW, Adusumalli S. Racial, Ethnic, and Socioeconomic Inequities in Glucagon-Like Peptide-1 Receptor Agonist Use Among Patients With Diabetes in the US. JAMA Health Forum. 2021 Dec 17;2(12):e214182. doi: 10.1001/jamahealthforum.2021.4182. eCollection 2021 Dec. PMID 35977298